CLINICAL TRIAL: NCT00000144
Title: Glaucoma Laser Trial (GLT) Glaucoma Laser Trial Followup Study (GLTFS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-43
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2006-06-05 (Estimated); Status verified 2003-10

CONDITIONS: Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

INTERVENTIONS:
Procedure: Argon Laser Treatment

SUMMARY:
To compare the safety and long-term efficacy of argon laser treatment of the trabecular meshwork with standard medical treatment for primary open-angle glaucoma.

DETAILED DESCRIPTION:
During the last decade, argon laser trabeculoplasty (ALT) has often been used instead of surgery as the treatment of choice in cases of open-angle glaucoma that could not be controlled by drugs. ALT treatment consists of tiny laser burns evenly spaced around the trabecular meshwork. It sometimes has been found to be effective in controlling glaucoma, although many eyes still require some medical treatment.

The Glaucoma Laser Trial (GLT), a randomized, controlled clinical trial, was conducted to determine whether ALT is effective in patients with newly diagnosed, primary, open-angle glaucoma. Each of the 271 patients in the trial received argon laser treatment in one eye and standard topical medication in the other eye. The eye to be started on medicine and the eye that would get the laser treatment were randomly selected. The Glaucoma Laser Trial Followup Study was a followup study of 203 of the 271 patients who enrolled in the Glaucoma Laser Trial. By the close of the Glaucoma Laser Trial Followup Study, median duration of followup since diagnosis of primary, open-angle glaucoma was 7 years (maximum, 9 years).

The argon laser treatment was done in two sessions 1 month apart, with one-half of the trabecular meshwork treated with 45 to 55 laser burns in each session. Patients were seen for a followup visit 3 months after the first laser treatment and every 3 months thereafter for a period of at least 2 years. At each visit, examination of the eyes included a check of intraocular pressure and visual acuity. Visual field examinations were performed 3, 6, and 12 months after randomization and annually thereafter. Disc stereo photographs were taken 6 and 12 months after randomization and annually thereafter.

The results of these examinations determined whether treatment should be changed. If the pressure in either eye had not been reduced to the desired level, the physician changed the medication in the eye treated with drops or started the use of drops in the laser-treated eye according to a standardized procedure being used in the trial. If intraocular pressure was still not successfully reduced, surgery or further laser treatment may have been required.

ELIGIBILITY:
At the time of recruitment, patients had to be at least 35 years old with an intraocular pressure of at least 22 mm Hg or greater in each eye and evidence of optic nerve damage in at least one eye.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1984-01

REFERENCES:
- [Background] The Glaucoma Laser Trial (GLT). 2. Results of argon laser trabeculoplasty versus topical medicines. The Glaucoma Laser Trial Research Group. Ophthalmology. 1990 Nov;97(11):1403-13. PMID 2255512
- [Background] The Glaucoma Laser Trial (GLT): 3. Design and methods. Glaucoma Laser Trial Research Group. Control Clin Trials. 1991 Aug;12(4):504-24. doi: 10.1016/0197-2456(91)90010-j. PMID 1657527
- [Background] The Glaucoma Laser Trial: 4. Contralateral effects of timolol on the intraocular pressure of eyes treated with ALT. GLT Research Group. Ophthalmic Surg. 1991 Jun;22(6):324-9. PMID 1896168
- [Background] The Glaucoma Laser Trial (GLT): 5. Subgroup differences at enrollment. Glaucoma Laser Trial Research Group. Ophthalmic Surg. 1993 Apr;24(4):232-40. PMID 8321504
- [Background] The Glaucoma Laser Trial (GLT): 6. Treatment group differences in visual field changes. Glaucoma Laser Trial Research Group. Am J Ophthalmol. 1995 Jul;120(1):10-22. doi: 10.1016/s0002-9394(14)73754-7. PMID 7611312
- [Background] The Glaucoma Laser Trial (GLT) and glaucoma laser trial follow-up study: 7. Results. Glaucoma Laser Trial Research Group. Am J Ophthalmol. 1995 Dec;120(6):718-31. doi: 10.1016/s0002-9394(14)72725-4. PMID 8540545
- [Background] The Glaucoma Laser Trial. I. Acute effects of argon laser trabeculoplasty on intraocular pressure. Glaucoma Laser Trial Research Group. Arch Ophthalmol. 1989 Aug;107(8):1135-42. PMID 2667508